CLINICAL TRIAL: NCT05714449
Title: OCT Eccentric Fixation, Fixation Stability, and Amblyopia in Children
Brief Title: OCT Eccentric Fixation and Amblyopia in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York College of Optometry (Other)
Responsible Party: Principal Investigator, Jingyun Wang, Associate Professor, State University of New York College of Optometry
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1912342
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Amblyopia
Keywords: eccentric fixation; amblyopia; patching; foveation therapy; OCT
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Patching group (Experimental): part-time patching following PEDIG guidelines.
  Interventions: Device: eye patch
- foveation therapy (Experimental): After-image foveation therapy training is 10 mins; MIT training is 5 minutes.
  Interventions: Device: After-image and MIT trainer

INTERVENTIONS:
Device: eye patch — standard amblyopia treatment
  Arms: Patching group
Device: After-image and MIT trainer — Common clinical training for foveation
  Arms: foveation therapy

SUMMARY:
The objectives of this proposal are to characterize the relationship between OCT eccentric fixation (OCT-EF), fixation eye movement (FEM), macular sensitivity in children with amblyopia.

DETAILED DESCRIPTION:
Aim 1. OCT EF changes with patching treatment at 12 weeks visit.

Aim 2. OCT EF changes with foveation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. children with best-corrected visual acuity (BCVA) of 20/40 (equivalent to 0.3 logMAR) or worse in the amblyopic eye (ranging from 20/40 to 20/400), and interocular difference of BCVA was at least two logMAR lines,
2. ocular causes of amblyopia that were identified as refractive(i.e., anisometropic, strabismus, or strabismic-anisometropic.

   * Anisometropia included interocular difference of spherical equivalent >=1D or interocular difference of astigmatism cylinder magnitude >=1D;
   * strabismus included those with deviation >=10PD or good alignment after prior strabismus surgery;
   * combined type included those who meet the criteria of both anisometropia and strabismus.
   * For the patching group, we will enroll 15 children with strabismic amblyopia who are prescribed patching treatment. Age: 4-12 years old.
   * For the foveation therapy group, we will enroll 15 children with strabismic amblyopia who are prescribed foveation therapies. Age: 8-16 years old.

Exclusion Criteria:

* born before 32 weeks gestational age;
* neurologic, developmental, or systemic illnesses known to be associated with ocular pathologies;
* congenital or acquired macular pathology.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-01-24 (Estimated); Study Completion 2026-01-24 (Estimated)

PRIMARY OUTCOMES:
OCT eccentric fixation | 12 weeks
  eccentric fixation measured with OCT imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Jingyun Wang, Principal Investigator — SUNY College of Optmetry
Locations (1):
- SUNY College of Optometry, New York, New York, United States